CLINICAL TRIAL: NCT05140564
Title: Safe Management of People With Type 1 Diabetes and EAting Disorders studY - Phase II
Brief Title: Safe Management of People With Type 1 Diabetes and EAting Disorders studY
Acronym: STEADY-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 290033
Record Dates: First submitted 2021-11-09; First posted 2021-12-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1; Eating Disorders
Keywords: Type 1 diabetes; Eating disorder; Diabulimia; EDNOS
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding and Eating Disorders; Diabulimia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEADY intervention group (Experimental)
  Interventions: Behavioral: STEADY intervention
- Treatment as usual group (control) (No Intervention)

INTERVENTIONS:
Behavioral: STEADY intervention — STEADY is a novel Cognitive Behavioural Therapy (CBT) based intervention for eating disorders in type 1 diabetes.
  Arms: STEADY intervention group

SUMMARY:
There is currently no effective intervention for type 1 diabetes and eating disorders. The main objective of STEADY Stage 2 is to test the feasibility of the newly developed STEADY intervention.

STEADY was co-designed by using Experience Based Co-Design methodology and other qualitative methods (focus groups, interviews).

These findings informed the development of a T1DM cognitive behaviour therapy (CBT) manual. The intervention will now be tested in a feasibility Randomised Controlled Trial (RCT) in adults with type 1 diabetes and eating disorders and compared with usual clinical care. If STEADY is feasible, this may provide an effective intervention for this population.

This study will take place at King's College London. Participants will remain in the study for 6 months, with a 12-month extended observation period. The study is expected to end in February 2023.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years);
2. Diagnosis of type 1 diabetes mellitus for at least 6 months;
3. Current disordered eating: defined as fear of insulin as weight gaining, avoidance/ restriction of insulin to control weight, food restriction, binge eating, any additional disordered eating behaviour as described by the 5th revision of the Diagnostic and Statistical Manual of Mental Disorders (DSM-V), or 11th Revision of the International Classification of Diseases (ICD-11); AND/OR score of 15 on EDE-QS, AND/OR a score of 20 on the DEPS-R.
4. Prepared to take part in a cognitive-behavioural therapy approach behaviour change strategy plus diabetes education intervention (with up to 12 sessions) with a varying proportion of face-to-face and virtual delivery mode;
5. Prepared to take part in the control group - treatment as usual (TAU)
6. Prepared to attend physical and mental health check-up at baseline and at the end of the intervention (control arm and intervention arm) face-to-face;
7. Currently under the care of a diabetes specialist team (as this study does not replace usual diabetes care);
8. Confirms availability to attend all sessions as part of the intervention (with the option of rescheduling sessions when necessary. Therapy sessions may be in person or via videoconference);
9. Investigator has confidence that the participant is able to fulfill all of the trial protocol requirements;
10. Participant has capacity to consent to the study. This is assessed by ability to explain information about their involvement in the study.

Exclusion Criteria:

1. HbA1c >15%/ 140.4 mmol/mol;
2. More than 2 admissions for DKA in the past 12 months;
3. More than 2 SH episodes (defined as needing 3rd party assistance) in the past 12 months due to insulin omission (not if triggered by infection or canula failure);
4. Severe mental illness, including severe depression with suicidal ideation, psychosis, emotionally unstable personality disorder requiring more intensive psychiatric treatment, substance problem use and dependence. (Potential participants with more severe mental illness are unlikely to benefit from a CBT based approach, therefore will be excluded to not delay their treatment. Investigators will use their clinical judgement, in agreement with the trial team. Mental health assessment by a psychiatrist is part of the baseline visit.);
5. Body mass index below 15kg/m2 or above 40kg/m2;
6. Significant cognitive impairment, e.g. dementia, learning disability;
7. Unable to speak/hear/understand/read/write in English;
8. Unable to give written informed consent;
9. Pregnant or planning pregnancy;
10. Advanced diabetes complications (end stage renal failure, registered blind, limb amputation);
11. Uncontrollable electrolyte disturbance, low blood pressure (<100/60mmHg), ECG abnormalities related to malnutrition (QTc-prolongation) or other physical conditions requiring inpatient treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months
  HbA1c measured in mmol/mol

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Stadler M, Zaremba N, Harrison A, Brown J, Pillay D, Allan J, Tan R, Ayis S, Konstantara E, Treasure J, Hopkins D, Ismail K. Safety of a co-designed cognitive behavioural therapy intervention for people with type 1 diabetes and eating disorders (STEADY): a feasibility randomised controlled trial. Lancet Reg Health Eur. 2025 Jan 20;50:101205. doi: 10.1016/j.lanepe.2024.101205. eCollection 2025 Mar. PMID 39902232